CLINICAL TRIAL: NCT05688384
Title: Patient-Controlled Sedation in Port Implantation (PACSPI-2) -a Randomized Controlled Trial
Brief Title: Patient-Controlled Sedation in Port Implantation (PACSPI-2)
Acronym: PACSPI-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Jönköping County (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT: 2021-003821-31
Record Dates: First submitted 2022-12-16; First posted 2023-01-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pain; Patient Satisfaction; Cancer; Venous Puncture
Keywords: patient-controlled sedation; totally implantable venous access device; subcutaneous implanted venous port; local anesthesia; propofol; alfentanil; indwelling catheter
MeSH Terms: conditions — Pain; Patient Satisfaction; Neoplasms | interventions — Propofol; Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (LA) (No Intervention): Patients in this arm will undergo SVP insertion in local anesthesia (LA)
- Study arm (LA+PCS) (Active Comparator): Patients in this arm will undergo SVP insertion in local anesthesia and PCS (LA+PCS)
  Interventions: Drug: Propofol + Alfentanil

INTERVENTIONS:
Drug: Propofol + Alfentanil — In addition to LA, patients in the study group are able to self-administer a combination of propofol and alfentanil using a patient-controlled sedation pump. The pump enables the patient via a hand-held button to trigger the release of a single bolus of 0.5ml containing 4.5mg propofol and 25µg alfentanil under an 10second period. This results in a maximal possible amount of 6 bolus doses per minute.
  Arms: Study arm (LA+PCS)

SUMMARY:
The goal of the study is to determine if patient-controlled sedation (PCS) with propofol and alfentanil reduces patient-reported pain perception during implantation of subcutaneous venous port (SVP).

The main question it aims to answer: How much pain did you (patient) experience during SVP-implantation Several other questions will be answered regarding: patient´s perception of the procedure, complication rate, procedure data.

The study contains two groups which will be compared. Control group: will do SVP implantation under local anaesthesia Study group: will do SVP implantation under local anaesthesia and patient-controlled sedation.

The patients are asked to complete a questionnaire postoperatively which contains questions on pain perception and satisfaction.

DETAILED DESCRIPTION:
The study is an open multicentre randomized controlled trial with a study and a control arm in a 1:1 ratio. Patients will be randomized to either a control arm of LA for SVP-implantation or a study arm of PCS with propofol and alfentanil as adjunct to LA for SVP-implantation. The aim is to randomize 340 patients with an estimated patient recruitment over 18 months with a following 6 months of data cleaning and analysis. The trial will be performed at two centres; County Hospital Ryhov, Jönköping, Sweden and University Hospital Linköping, Sweden. SVP implantation procedure and perioperative time period is estimated to 2-4 hours. The primary endpoint is assessment of patients´ self-reported pain perception. Secondary outcomes include patient satisfaction, implantation conditions, sedation level, sedative and analgesic medication consumption, procedural time consumption as well as safety aspects, adverse events and estimation of perioperative experience. Participation in the trial ends after telephone inquiry one day postoperatively.

Control arm:

SVP-implantation in LA:

Subcutanous venous ports were introduced in 1981. A SVP is a small device around 3cm in diameter with an injectable membrane buried just under the skin. It is connected to a thin tube with its tip in a large bore vein. Access to the SVP is achieved by puncturing the skin with a needle.

Local anaesthetic causes the absence of pain sensation in the location where applied by decreasing the rate of depolarization and repolarization of excitable membranes such as nociceptors and nerves. The most commonly used solutions are from the amide group differing in pharmacokinetics. In order to reduce a burning sensation on infiltration substances can be combined with sodium bicarbonate. There will be no restrictions in the choice of LA-solution being left up to local practice at participating sites. With the beginning of the procedure LA is subcutaneously applied to patients in both groups. LA used at participating centres are Mepivacaine 10mg/ml, 20-40ml subcutaneously or Lidnocaine 10mg/ml, 20-40 ml subcutaneously.

Study arm:

SVP-implantation in LA and PCS:

In addition to LA, patients in the study group are able to self-administer a combination of propofol and alfentanil using a patient-controlled sedation pump. The pump enables the patient via a hand-held button to trigger the release of a single bolus of 0.5ml containing 4.5mg propofol and 25µg alfentanil under an 10 second period. This results in a maximal possible amount of 6 bolus doses per minute.

Propofol is a short-acting anaesthetic agent commonly used for general anaesthesia and procedural sedation. Several mechanisms of action have been proposed both through potentiation of GABAA receptor activity and in higher doses behaving as GABAA receptor agonist. When used for intravenous sedation a single dose wears off within minutes demanding for continuous or intermittent application.

Alfentanil is a short-acting synthetic opioid analgesic agent with rapid onset of effects at µ-opioid receptors. These properties make it suitable to provide analgesia for brief procedures and to infuse for longer procedures and yet provide relatively rapid recovery.

Rescue sedation will be available to patients in both groups on the patient´s or operator´s demand. Rescue sedation consists of propofol and alfentanil administered by the clinician and is documented in the e-CRF.

Setting:

This trial will be carried out in the following anaesthesia departments:

OP/IVA clinic, County Hospital Ryhov, Sweden AnOpIVA clinic, University Hospital Linköping, Sweden

Participants will be instructed on use of the PCS pump (Syramed µSP6000, Arcomed AG, Switzerland) by a nurse anesthetist. The syringe is loaded with 36 ml propofol (10 mg/ml) and 4 ml alfentanil (0.5 mg/ml). Each time the patient presses the handheld button, an aliquot of 0.5 ml is injected (4.5 mg propofol/0.025 mg alfentanil). The injection time is set to 10 s, restricting self-administration to a maximum of 6 bolus doses per minute corresponding to 27 mg propofol and 0.15 mg alfentanil per minute. No lockout period is applied. Local anaesthesia is injected in the operating site. Vital parameters prior to the procedure are recorded. Patients are monitored using electrocardiography for heartrate (HR), non-invasive blood pressure (BP), oxygen saturation (SpO2), and respiratory rate (RR) at 5-min intervals during the procedure. Bradycardia is defined as HR <40 beats/min, tachycardia as HR >100 beats/min, hypotension as systolic BP < 90 mmHg or a decrease of >30% from baseline, hypoxia as SpO2 <90% or a decrease of >5% from baseline, and bradypnea as RR of <8 breaths per minute. Supplemental oxygen via a capnograph-fitted nasal cannula is administered to all patients at 2 L/min during the procedure. The Observer's Assessment of Alertness/Sedation score (OAA/S) [9] is used to determine the sedation level during the four procedural steps: 1) sterile swabbing, 2) injection of LA, 3) catheter tunneling, and 4) sterile drape removal. The operating anesthesiologist assesses the operating conditions on a 4 point scale with 1 enabling the operator to perform the procedure without time delay and 4 having to abort the procedure. Puncture attempt is defined as continuous needle advancement to establish vein puncture. An unvalidated patient perception assessment tool with seven dimensions applying the NRS is used to evaluate patient perception. QoR-15 will be measured att 3 timepoints. Preoperatively, postoperatively before patient discharge and one day postoperatively.

QoR- 15 data sampling was planned a priori to the trial start of PACSPI 2. QoR-15 data was listed as secondary outcome in the protocol and on clinicaltrials.gov. After study commencement we became aware of the importance of not only reporting overall QoR-15 score but even recovery time trajectories for the separate time periods within the allocated groups. Moreover, since QoR-15 is a composite score, positive scores in some domains may be counterbalanced by negative scores in other domains, therefore reporting an aggregate score may cause loss of potentially important, more granular data. To specifically address these questions, we will conduct a pre-planned substudy addressing the trajectories of recovery and domain by domain changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with cancer in need of SVP.

Exclusion Criteria:

* Inability to operate the PCS apparatus.

  * Inability to communicate in Scandinavian languages.
  * Patients who require general anaesthesia or patients eligible for LA only on anesthesiologist´s assessment (i.e. severe sleep apnea).
  * Propofol or alfentanil allergy.
  * Non-fasting according to guidelines of the Swedish Society for Anaesthesia and Intensive Care (SFAI).
  * Failure to achieve peripheral vascular access.
  * Pregnancy
  * Previous participation in study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Maximal intraprocedural pain level on numeric rating scale | after completion of procedure 10 minutes before discharge
  NRS Participants assessment of maximal pain level experienced during the procedure using a numeric rating scale from 0-10 (0=no pain, 10=worst pain I know) on patient questionnaire.

SECONDARY OUTCOMES:
Participants overall satisfaction, Participants satisfaction with staff | after completion of procedure 10 minutes before discharge
  NRS Participants assessment of overall satisfaction experienced during the procedure using a numeric rating scale from 0-10 (0=not satisfied at all, 10=very satisfied) on patient questionnaire
Number of participants with arterial puncture, pneumothorax, bradycardia, hypoxia, airway intervention, bradypnea | during the procedure
  Respiratory and circulatory complications as well as mechanical complications during the procedure bradycardia: defined as heart < 40/minutes during the procedure Hypoxia: defined as Oxygen saturation <90% or significant drop from baseline (>5% SaO2 drop) during the procedure Airway intervention: defined as intervention by staff with chin lift during the procedure bradypnea: defined as respiratory rate <8/minute during the procedure
Sedation score on Observers Assessment of Alertness/Sedation scale (OAA/S) | during procedure at time point T1: sterile skin prepping; T2: local anaesthetic injection; T3: tunneling procedure; T4: draping removal
  Sedation levels according to Observers Assessment of Alertness/Sedation scale 5: responds readily to naame spoken in normal tone 4: responds lethargically to name spoken in normal tone 3: responds only after name is called loudly, repeatedly, or both 2: responds only after mild prodding or shaking
  1: responds only after painful trapezius squeeze 0: does not respond to painful trapezius squeeze
type of catheter | during the procedure
  Procedural measures
amount and type of local anaesthesia | during the procedure
  Procedural measures
amount of sedative medication given | during the procedure
  Procedural measures
time consumption of the procedure | during the procedure
  Procedural measures
number of puncture attempts | during the procedure
  Procedural measures
use of ultrasound | during the procedure
  Procedural measures
positioning of catheter tip | during the procedure
  Procedural measures
vessel choice | during the procedure
  Procedural measures
Quality of Recovery QoR-15 questionnaire | by telephone the day after the procedure
  Quality of Recovery according to QoR-15 Have you had any of the following in the last 24 hours? 10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor])
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal
  6. Able to communicate with family or friends
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed
Quality of Recovery QoR-15 questionnaire | before the procedure at arrival to preoperative unit
  Quality of Recovery according to QoR-15
Quality of Recovery QoR-15 questionnaire | within 1 hour after completion of procedure
  Quality of Recovery according to QoR-15
Participants evaluation of the importance of receiving sedatives during the procedure Participants evaluation of the importance of being in control of sedation administration | within 1 hour after completion of procedure
  Participants assessment of the importance of receiving sedatives and being in control of sedation on a numeric rating scale from 0-10 (0=not important, 10=very important) on patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Seifert, Principal Investigator — Region Jönköping
Locations (1):
- Länssjukhuset Ryhov, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for sharing on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The supporting information will be available from november 2022.
Access Criteria: Requests for sharing IPD that underlie results in a publication can be made to the principal investigator.
  The supporting information will be available on researchgate.com.

REFERENCES:
- [Background] Taxbro K, Hammarskjold F, Thelin B, Lewin F, Hagman H, Hanberger H, Berg S. Clinical impact of peripherally inserted central catheters vs implanted port catheters in patients with cancer: an open-label, randomised, two-centre trial. Br J Anaesth. 2019 Jun;122(6):734-741. doi: 10.1016/j.bja.2019.01.038. Epub 2019 Apr 17. PMID 31005243
- [Background] Grossmann B, Nilsson A, Sjoberg F, Bernfort L, Nilsson L. Patient-controlled sedation with propofol for endoscopic procedures-A cost analysis. Acta Anaesthesiol Scand. 2020 Jan;64(1):53-62. doi: 10.1111/aas.13463. Epub 2019 Oct 10. PMID 31436310
- [Background] Kreienbuhl L, Elia N, Pfeil-Beun E, Walder B, Tramer MR. Patient-Controlled Versus Clinician-Controlled Sedation With Propofol: Systematic Review and Meta-analysis With Trial Sequential Analyses. Anesth Analg. 2018 Oct;127(4):873-880. doi: 10.1213/ANE.0000000000003361. PMID 29750696
- [Background] Clements W, Sneddon D, Kavnoudias H, Joseph T, Goh GS, Koukounaras J, Snow T. Randomized and controlled study comparing patient controlled and radiologist controlled intra-procedural conscious sedation, using midazolam and fentanyl, for patients undergoing insertion of a central venous line. J Med Imaging Radiat Oncol. 2018 Dec;62(6):781-788. doi: 10.1111/1754-9485.12817. Epub 2018 Oct 8. PMID 30295410
- [Background] Burlacu CL, McKeating K, McShane AJ. Remifentanil for the insertion and removal of long-term central venous access during monitored anesthesia care. J Clin Anesth. 2011 Jun;23(4):286-91. doi: 10.1016/j.jclinane.2010.12.007. PMID 21663812
- [Derived] Seifert S, Taxbro K, Nilsson A, Azman J, Chew MS, Hammarskjold F. Patient-Controlled Sedation in Port Implantation (PACSPI 2)-A Randomised Clinical Trial. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70148. doi: 10.1111/aas.70148. PMID 41214479

DOCUMENTS (2):
  • Study Protocol (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT05688384/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT05688384/SAP_000.pdf